CLINICAL TRIAL: NCT02070770
Title: The Effect of Short-term Adherence to a Very Low Calorie Diet on Heart Rate Variability: a Pilot Randomised Controlled Trial in Obese Men and Women
Brief Title: The Effect of a Short-term Very Low Calorie Diet on Heart Rate Variability in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Lighterlife Ltd (UK) (Unknown)
Responsible Party: Principal Investigator, Dr Wendy Hall, Lecturer in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LHS2014
Record Dates: First submitted 2014-02-23; First posted 2014-02-25 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very low calorie diet (Experimental)
  Interventions: Dietary Supplement: Very low calorie diet
- Standard weight loss diet (Active Comparator)
  Interventions: Other: Standard weight loss diet

INTERVENTIONS:
Dietary Supplement: Very low calorie diet
  Other Names: Lighterlife Total
  Arms: Very low calorie diet
Other: Standard weight loss diet
  Arms: Standard weight loss diet

SUMMARY:
The purpose of this study is to determine whether short-term adherence to a very low calorie diet is effective in improving heart rate variability in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking men and women
* Aged 32-65 years
* BMI 30-42 kg/m2

Exclusion Criteria:

* History of cardiovascular disease, diabetes, cancer, renal or liver disease or chronic gastrointestinal disorder
* Epileptic or history of fainting
* Adhered to a VLCD in the past 6 months
* History of drug or alcohol abuse including heavy drinking.
* Pregnancy, planning to get pregnant or breastfeeding
* Currently taking medications to control blood pressure
* Weight change of over 3kg in the past two months

Ages: 32 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 24 h SDNN (mean of the standard deviations of the normal-to-normal intervals) at day 7 | Baseline, day 7
  SDNN is a time domain parameter of overall heart rate variability

SECONDARY OUTCOMES:
Change from baseline in night-time SDNN (mean of the standard deviations of the normal-to-normal intervals) at day 7 | Baseline, day 7
Change from baseline in daytime SDNN (mean of the standard deviations of the normal-to-normal intervals) at day 7 | Baseline, day 7
Change from baseline in 24 h mean IBI (interbeat interval) at day 7 | Baseline, day 7
Change from baseline in night-time mean IBI (interbeat interval) at day 7 | Baseline, day 7
Change from baseline in daytime mean IBI (interbeat interval) at day 7 | Baseline, day 7
Change from baseline in 24 h SDANN (standard deviations of the average normal-to-normal intervals calculated over periods of 5-minutes) at day 7 | Baseline, day 7
Change from baseline in night-time SDANN (standard deviations of the average normal-to-normal intervals calculated over periods of 5-minutes) at day 7 | Baseline, day 7
Change from baseline in daytime SDANN (standard deviations of the average normal-to-normal intervals calculated over periods of 5-minutes) at day 7 | Baseline, day 7
Change from baseline in 24 h triangular index at day 7 | Baseline, day 7
Change from baseline in night-time triangular index at day 7 | Baseline, day 7
Change from baseline in daytime triangular index at day 7 | Baseline, day 7
Change from baseline in 24 h RMSSD (root mean square of successive differences of normal-to-normal differences) at day 7 | Baseline, day 7
Change from baseline in night-time RMSSD (root mean square of successive differences of normal-to-normal differences) at day 7 | Baseline, day 7
Change from baseline in daytime RMSSD (root mean square of successive differences of normal-to-normal differences) at day 7 | Baseline, day 7
Change from baseline in 24 h pNN50 (% differences between adjacent normal-to-normal intervals that are >50 ms) at day 7 | Baseline, day 7
Change from baseline in night-time pNN50 (% differences between adjacent normal-to-normal intervals that are >50 ms) at day 7 | Baseline, day 7
Change from baseline in daytime pNN50 (% differences between adjacent normal-to-normal intervals that are >50 ms) at day 7 | Baseline, day 7
Change from baseline in 24 h LF (low frequency power) at day 7 | Baseline, day 7
Change from baseline in night-time LF (low frequency power) at day 7 | Baseline, day 7
Change from baseline in daytime LF (low frequency power) at day 7 | Baseline, day 7
Change from baseline in 24 h HF (high frequency power) at day 7 | Baseline, day 7
Change from baseline in night-time HF (high frequency power) at day 7 | Baseline, day 7
Change from baseline in daytime HF (high frequency power) at day 7 | Baseline, day 7
Change from baseline in 24 h LF/HF at day 7 | Baseline, day 7
Change from baseline in night-time LF/HF at day 7 | Baseline, day 7
Change from baseline in daytime LF/HF at day 7 | Baseline, day 7
Change from baseline in 24 h VLF (very low frequency power) at day 7 | Baseline, day 7
Change from baseline in night-time VLF (very low frequency power) at day 7 | Baseline, day 7
Change from baseline in daytime VLF (very low frequency power) at day 7 | Baseline, day 7

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Hall, PhD, Principal Investigator — King's College London
Locations (1):
- Diabetes & Nutritional Sciences Division, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] F Fitzpatrick, A White, R Allen, A Pinto & W Hall. Short-term adherence to a very low calorie diet increases heart rate variability and reduces 24 hours heart rate in obese subjects: a randomised controlled pilot study. Journal of Human Nutrition and Dietetics. 2016; 29 (Suppl. 1), 45-46, AB47.